CLINICAL TRIAL: NCT05848960
Title: Nutritional Support With Mediterranean Diet and Hyper Caloric, Hyperproteic Oral Supplements in Heart Failure Sarcopenia
Brief Title: Mediterranean Diet and Nutritional Support in Heart Failure Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Heart failure sarcopenia 1
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
Keywords: Heart failure; Sarcopenia; Nutritional support
MeSH Terms: conditions — Sarcopenia; Heart Failure | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mediterranean diet (Active Comparator): Mediterranean diet
  Interventions: Other: Mediterranean diet
- Mediterranean diet plus hypercaloric, hyperproteic oral supplement (Experimental): Mediterranean diet plus hypercaloric, hyperproteic oral supplement
  Interventions: Dietary Supplement: Hypercaloric, hyperproteic oral supplement; Other: Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Hypercaloric, hyperproteic oral supplement — 2 supplements per day
  Arms: Mediterranean diet plus hypercaloric, hyperproteic oral supplement
Other: Mediterranean diet — Mediterranean diet

SUMMARY:
Heart failure (HF) is a chronic disease with an increasing incidence; it represents the final stage of multiple cardiac diseases and significantly affects the QoL of the patients. Its prevalence is about 26 million people in the world, especially in elderly. Sarcopenia has been directly associated with the presence of increased comorbidity in patients with HF. In this study the investigators aim to compare the clinical evolution of patients with HF after receiving nutritional support with Mediterranean diet alone or in combination with a hypercaloric, hyperproteic oral nutritional Supplement

DETAILED DESCRIPTION:
All participants will receive general counseling, education about MedDiet and vitamin D supplementation in order to reach levels of sufficiency (25OH vitamin D>30 ng/dL) for avoiding confounding results. Participants (n=50) will be randomly allocated to MedDiet or MedDiet plus hypercaloric, hyperproteic standard oral nutritional supplement (ONS), 2 ONS per da). Participants will be evaluated at baseline, 12 and 24 weeks after nutritional support

ELIGIBILITY:
Inclusion Criteria:

* - Patients with a previous admission due to HF in the previous 12 months
* Moderate or severe LVEF
* Both sexs
* Age >18 years old.

Exclusion Criteria:

* MDRD <15 ml/min
* End-stage liver disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 6 months
  Changes in percent of muscle mass
Left ventricular ejection fraction | 6 months
  Changes in left ventricular ejection fraction

SECONDARY OUTCOMES:
pro-BNP | 6 months
  Changes in pro-BNP
Fat mass | 6 months
  Changes in fat mass using bioimpedance and echography
Phase angle | 6 months
  Changes in phase angle using bioimpedance
Albumin | 6 months
  Changes in serum albumin levels (g/l)
Preallbumin | 6 months
  Changes in serum prealbumin levels (mg/dl)
Transferrin | 6 months
  Changes in serum transferrin levels (mg/dl)
CRP | 6 months
  Changes in CRP levels (g/l)

CONTACTS AND LOCATIONS:
Locations (1):
- IMIBIC, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No